CLINICAL TRIAL: NCT03799887
Title: Effects of Different Percentages Body Weight Supported Treadmill Training on Gait, Balance, Quality of Life and Fatigue in Parkinson's Disease: A Double Blind Randomized Controlled Trial
Brief Title: Effects of Different Percentages Body Weight Supported Treadmill Training on Gait, Balance, Quality of Life and Fatigue in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Tuğba Atan, Assoc. Prof., Hitit University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-171
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; gait; balance; treadmill training; fatigue
MeSH Terms: conditions — Parkinson Disease; Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0% unweighed BWSTT (Active Comparator): 0% unweighed Body Weight Supported Treadmill Training
  Interventions: Behavioral: 0% unweighed BWSTT
- 10% unweighed BWSTT (Experimental): 0% unweighed Body Weight Supported Treadmill Training
  Interventions: Behavioral: 10% unweighed BWSTT
- 20% unweighed BWSTT (Experimental): 20% unweighed Body Weight Supported Treadmill Training
  Interventions: Behavioral: 20% unweighed BWSTT

INTERVENTIONS:
Behavioral: 0% unweighed BWSTT — 30 minutes conventional rehabilitation program (CRP) including range of motion, stretching and strengthening exercises for upper and lower extremities, balance and mobility exercises.
  After CRP, participants were provided 30 minutes 0% unweighed BWSTT sessions including a 5 minutes warm - up and cool - down period for each session, 5 days a week, for 6 weeks (totally, 30 sessions).
  Arms: 0% unweighed BWSTT
Behavioral: 10% unweighed BWSTT — 30 minutes conventional rehabilitation program (CRP) including range of motion, stretching and strengthening exercises for upper and lower extremities, balance and mobility exercises.
  After CRP, participants were provided 30 minutes 10% unweighed BWSTT sessions including a 5 minutes warm - up and cool - down period for each session, 5 days a week, for 6 weeks (totally, 30 sessions).
  Arms: 10% unweighed BWSTT
Behavioral: 20% unweighed BWSTT — 30 minutes conventional rehabilitation program (CRP) including range of motion, stretching and strengthening exercises for upper and lower extremities, balance and mobility exercises.
  After CRP, participants were provided 30 minutes 20% unweighed BWSTT sessions including a 5 minutes warm - up and cool - down period for each session, 5 days a week, for 6 weeks (totally, 30 sessions).
  Arms: 20% unweighed BWSTT

SUMMARY:
Body weight supported treadmill training (BWSTT) is an important rehabilitative choice for neurologically impaired subjects such as Parkinson's disease (PD). The aim of the study is to evaluate the effectiveness of different percentages BWSTT on gait, balance, quality of life and fatigue in moderate to advanced PD.

DETAILED DESCRIPTION:
Body weight supported treadmill training (BWSTT) is an important rehabilitative choice for neurologically impaired subjects such as Parkinson's disease (PD). The aim of the study is to evaluate the effectiveness of different percentages BWSTT on gait, balance, quality of life and fatigue in moderate to advanced PD. Thirty five patients were randomly assigned to one of the three groups according to the percentage unweighed: 0% BWSTT, 10% BWSTT and 20% BWSTT. All patients participated 30 minutes BWSTT sessions 5 days a week, for 6 weeks. Primary outcomes were 6 minute walk test (6MWT), Berg balance scale (BBS), Unified Parkinson's Disease Rating Scale (UPDRS); and secondary outcomes were Nottingham health profile (NHP), Fatigue Impact Scale (FIS) and Fatigue Severity Scale (FSS) which were performed at the beginning and end of the rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's disease according to the UK Brain Bank criteria.
* Subjects had clinically moderate to advanced severity of disease (Hoehn and Yahr stage 2 - 4).
* Subjects whose medical treatment had been on stable dosage of dopaminomimetics for at least 4 weeks before the study.
* Subjects ability to walk with or without assistive device.

Exclusion Criteria:

* Subjects had cardiovascular, inflammatory or musculoskeletal problems that could prevent them to participate in an exercise program.
* Subjects whose mini mental status examination score was less than 26.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-10-20 (Actual); Primary Completion 2010-10-20 (Actual); Study Completion 2012-11-20 (Actual)

PRIMARY OUTCOMES:
6 Minute Walk Test (6MWT) | 6 weeks
  Functional exercise capacity was assessed by distance walked in 6 minutes (6MWT). The patient was asked to walk as long as possible for 6 minutes on a 30 meters of marked and flat ground, at a self selected speed. 6MWT is a submaximal exercise test and can be used to assess treatment response .
Berg Balance Scale (BBS): | 6 weeks
  It contains 14 instructions and 0 - 4 points is given for each instruction according to the performance of the patients. 0 points are given when the patient totally could not do the activity while 4 points are given when the patient completes the activity independently.
Unified Parkinson's Disease Rating Scale (UPDRS): | 6 weeks
  It is used to follow the clinical status of PD. It consists of four main parts (totally 183 points): mentation, behavior and mood (UPDRS I: 16 points), activities of daily living (UPDRS II: 52 points), motor examination (UPDRS III: 92 points), treatment complications (UPDRS IV: 23 points).

SECONDARY OUTCOMES:
Nottingham Health Profile (NHP): | 6 weeks
  It contains 38 items that address pain, physical mobility, emotional reactions, energy, social isolation, and sleep dimensions. Higher scores indicate worse quality of life.
Fatigue Impact Scale (FIS): | 6 weeks
  This scale assesses the cognitive, physical and social effects of fatigue during the last one week in a total of 40 - item questionnaire (0 = no problem, 4 = maximum problem).
Fatigue Severity Scale (FSS): | 6 weeks
  This scale assesses the severity of fatigue during the last one week in a total of 9 - item questionnaire (1 = strongly disagree, 7 = strongly agree). The total score ranges from 9 - 63, in which higher score means higher severity of fatigue .

CONTACTS AND LOCATIONS:
Locations (1):
- Tuğba Atan, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes